CLINICAL TRIAL: NCT02447471
Title: Agreement of the Nexfin™ Non-invasive Cardiac Output Monitor With Non-invasive Blood Pressure Measurement in Patients Undergoing Cesarean Delivery Under Spinal Anesthesia: a Pilot Observational Study
Brief Title: Agreement of the Nexfin™ Monitor With Non-invasive Blood Pressure Measurement
Acronym: Nexfin Pilot
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: H15-00992
Record Dates: First submitted 2015-05-14; First posted 2015-05-18 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Blood Pressure Measurement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- study group: all participants
  Interventions: Device: Nexfin

INTERVENTIONS:
Device: Nexfin — Nexfin cuff placed on finger to measure blood pressure

SUMMARY:
Currently, BP is measured using an inflatable cuff wrapped around the patient's upper arm. This can be set to inflate every minute, but measurement may fail due to patient movement or shivering. Failed measurement occurs in up to 38% of patients.

This study aims to determine how the Nexfin device - which measures BP using a cuff wrapped around a finger - compares to standard BP measurement.

DETAILED DESCRIPTION:
This study aims to determine how the Nexfin device - which measures BP using a cuff wrapped around a finger - compares to standard BP measurement.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female pregnant patients
* ≥19 years old
* Undergoing elective Cesarean section under spinal or combined spinal-epidural anesthesia

Exclusion Criteria:

* Contraindication to wearing Nexfin cuff (upper limb vascular disease, amputated digits)
* Obesity (BMI > 38 kg/m2)
* Use of arterial line for BP measurement
* Inability to read and understand English

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: BC Women's hospital parturients
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-05; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Nexfin bp vs NIBP | During cesarean delivery

CONTACTS AND LOCATIONS:
Overall Officials: Vit Gunka, MD FRCPC, Principal Investigator — University of British Columbia
Locations (1):
- BC Women's Hospital, Vancouver, British Columbia, Canada